CLINICAL TRIAL: NCT03135496
Title: Evaluation of Endothelial Dysfunction During Aortic Valvular Replacement by Bioprosthesis With and Without Extracorporeal Circulation
Acronym: DYVA2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2016_843_0029
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Endothelial Dysfunction; Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery with CEC
  Interventions: Other: Study of endothelial function biological markers
- Without CEC
  Interventions: Other: Study of endothelial function biological markers

INTERVENTIONS:
Other: Study of endothelial function biological markers — Study of endothelial function biological markers

SUMMARY:
Patients with aortic stenosis present many risk factors for endothelial dysfunction (arterial hypertension, arteriosclerosis, dyslipidemia, chronic renal insufficiency, etc.). It is likely that a significant number of patients suffer from pre-existing endothelial dysfunction that can be evaluated by a molecular approach.

To date, the replacement of the aortic valve can be performed by surgery with extracorporeal circulation (CEC) or percutaneous (Transcatheter Aortic Valve ImplantationTAVI) without CEC.

Two recent studies have demonstrated a sustained improvement in endothelial function with TAVI. On the contrary, studies have demonstrated that post-operative complications (coagulopathy, capillary leak syndrome, acute vasoplastic disorder and acute renal failure) after surgery with extracorporeal circulation (CEC) could be the result of the interaction between pre-existing endothelial dysfunction And the "operative" aggression associated with the CEC.

Thus, patients with preexisting involvement of endothelial function would develop vascular dysfunction after valvular replacement due to "endothelial activation" related to CEC. This phenomenon would not exist in TAVI, and would explain the absence of so-called vascular dysfunction complications (Systemic inflammatory response syndrome, vasoplastic syndrome, disseminated intravascular coagulation).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years.
* Patient operated on aortic valvular replacement by bioprosthesis in surgery + CEC or TAVI
* Signed consent.
* Affiliation to Social Security

Exclusion Criteria:

* Any other cardiac surgery
* Mechanical aortic valve replacement
* Permanent Ac / Fa.
* Pregnant woman.
* Curative anticoagulation (AVK, NANCO, heparin).
* Patient under tutelage or curatelle.
* Refusal of the patient.
* Participation in another study.
* Preoperative sepsis
* Minor or adult, under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (Angiopoietin 1 and 2) in two types of populations: one with CEC and one without CEC (TAVI).
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Analysis of the variation of the following endothelial function markers: angiopoetin 1 and 2 depending on whether or not extracorporeal circulation | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France